CLINICAL TRIAL: NCT03580642
Title: Efficacy and Usability of eHealth Technologies in Stroke Survivors for Prevention of a New Stroke and Improvement of Self-management: Phase III Randomized Control Trial
Brief Title: Decision Support System for Stroke Survivors
Acronym: STARR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biobizkaia Health Research Institute (Other Government)
Responsible Party: Principal Investigator, Leire Ortiz Fernández, Principal Investigator, Biobizkaia Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STARR
Record Dates: First submitted 2017-12-22; First posted 2018-07-09 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Telerehabilitation; Stroke; Life Style
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: We will perform a randomised, pilot, prospective, parallel group, open, and unicentric Clinical Trial (RCT) with stroke survivors and their caregivers at Cruces University Hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eHealth Technologies (Experimental): eHealth Technologies is a messure of diferent paramenters of the patient; heart rate, blood pressure, weight, thermometer, daily activity.
  Interventions: Device: eHealth Technologies
- Control (No Intervention): Habitual treatment.

INTERVENTIONS:
Device: eHealth Technologies — The controls will get a conventional treatment from the acute to the chronic phase of stroke and the cases will get a conventional treatment till the end of the subacute phase. However, in the chronic period they will use the developed STARR App and DSS, as well as commercial wearables.
  Arms: eHealth Technologies

SUMMARY:
The aim of the study is to evaluate the usability of the system and its accordance with the users' needs. This evaluation will consider the effectiveness and the efficiency of the system, as well as stroke survivors' satisfaction. The effectiveness and the efficiency of the system will be measured by:

* The relationship between the control of stroke survivors' daily activities and their risk of having a secondary stroke,
* The decrease of the need for caregivers,
* And consequently an improvement in stroke survivors' self-management.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the usability of the system and its accordance with the users' needs. This evaluation will consider the effectiveness and the efficiency of the system, as well as stroke survivors' satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years.
* First ischemic stroke within the past 6 months.
* Hemiparesia with mild (91-99)-moderate (61-90) disability (Barthel Index).
* With or without speech patology but able to understand simple orders ( >45).
* Able to cope and to understand the guidelines to use the devices.
* Informed consent signed.

Exclusion Criteria:

* Life expectancy <12 months.
* Severe cognitive impairments.
* Medical comorbidities that could interfere with the home-rehabilitation program (MoCA < 26).
* Socio-familiar dystocia (SFES ≥ 14).
* Modified Rankin Scale > 1.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-27 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale | 12 months
  The System Usability Scale (SUS) provides a "quick and dirty", reliable tool for measuring the usability.
  Developers work to create systems that are easy and straight-forward for people to use. Terms such as "user friendly" and "easy-to-use" often indicate these characteristics, but the overall technical name for them is usability.

SECONDARY OUTCOMES:
Age | 12 months
  This an outcome to evaluate the eligibility of the patient. Age variable will be in years.
Stroke date | 12 months
  This an outcome to evaluate the eligibility of the patient. This variable will be the patient stroke date.
Oxfordshire Community Stroke Project Classification | 12 months
  This an outcome to evaluate the eligibility of the patient. This variable will be useful in estimation of after stroke complications and prognostication.
Modified Barthel Index | 12 months
  This an outcome to evaluate the eligibility of the patient. This variable will assessing self care and mobility activities of daily living of the patient.
Mississippi Aphasia Screening Test | 12 months
  This an outcome to evaluate the eligibility of the patient. This variable will to be used to detect changes in language abilities over time of the patient.
Montreal Cognitive Assessment | 12 months
  This an outcome to evaluate the eligibility of the patient. This variable will be collected for detecting cognitive impairment of the patient.
Gijon's social-familial evaluation Scale | 12 months
  Assess the social and family situation of people living in the home. Detect risk situations and social problems.
  There are no subscales. It has a global score. Score between 0-20 points, indicating higher score worse social situation.
Charlson Comorbidity Index | 12 months
  This an outcome to evaluate the eligibility of the patient.
Gender | 12 months
  This is a socio demographic outcome. This outcome will be collected as Male or Female.
Ethnic group | 12 months
  This is a socio demographic outcome.
Deprivation index | 12 months
  This is a socio demographic outcome.
Hand dominance | 12 months
  This is a socio demographic outcome. This outcome will be collected as right-handed and left-handed.
Education level | 12 months
  This is a socio demographic outcome.
Type of profession | 12 months
  This is a socio demographic outcome.
Hobbies | 12 months
  This is a socio demographic outcome.
Medical Research Council Scale | 12 months
  Scale for testing muscle strength in palsy. There are no subscales. It measures from Grade 0 (No contraction) to Grade 5 (Normal strength).
MAST Test | 12 months
  This is a neurological physical examination.
MoCA Test | 12 months
  This is a neurological physical examination.
Functional Ambulation Categories | 12 months
  This is a neurological physical examination.
10 Meters Walking Test | 12 months
  This is a neurological physical examination. The variable will collected in m/sg.
6 Minutes Walking Test | 12 months
  This is a neurological physical examination. The variable will collected in metres.
Berg Balance Scale | 12 months
  This is a neurological physical examination.
Frenchay Arm Test | 12 months
  This is a neurological physical examination.
Asworth Modified Scale | 12 months
  Scale for testing muscle spasticity. It rates severity of tone. There are no subscales. It measures from Grade 0 (No increase in muscle tone) to Grade 4 (Affected part(s) rigid in flexion or extension).
Fatigue Severity Scale | 12 months
  To measure the fatigue caused by a number of chronic medical conditions. There are no subscales. It has a global score. The FSS questionnaire contains nine statements. A low value (e.g., 1) indicates strong disagreement with the statement, whereas a high value (e.g., 7) indicates strong agreement. The total mean score is 7 points. FSS mean score > 4 indicates severe fatigue.
Line Bisection Test | 12 months
  This is a neurological physical examination.
Disphagia | 12 months
  This is a neurological physical examination.
Campimetry | 12 months
  This is a neurological physical examination.
Analogic Visual Scale | 12 months
  This is a neurological physical examination.
Analgesic Treatments | 12 months
  This is a neurological physical examination.
Golberg Scale | 12 months
  This is a cardiovascular risk factor. To messure depression and anxiety.
Weight | 12 months
  This is a cardiovascular risk factor. In kg
Height | 12 months
  This is a cardiovascular risk factor. In meter
BMI | 12 months
  This is a cardiovascular risk factor.
Waist Size | 12 months
  This is a cardiovascular risk factor.
Waist to Hip Ratio | 12 months
  This is a cardiovascular risk factor.
Blood Pressure | 12 months
  This is a cardiovascular risk factor. In mmHg
Heart Rate | 12 months
  This is a cardiovascular risk factor.
Glycaemia | 12 months
  This is a cardiovascular risk factor.
Health Literacy Test | 12 months
  This is for measure the health literacy of the patient.
Mediterranean Diet Assessment Test | 12 months
  This is for measure the life style of the patient.
Physical Activity | 12 months
  This is for measure the life style of the patient.
Toxic Consumption | 12 months
  This is for measure the life style of the patient.
Total Cholesterol | 12 months
  This is a blood test for measure the lipidic profile of the patient.
HDL | 12 months
  This is a blood test for measure the lipidic profile of the patient.
LDL | 12 months
  This is a blood test for measure the lipidic profile of the patient.
Proteins | 12 months
  This is a blood test of the patient.
Albumin | 12 months
  This is a blood test of the patient.
HbA1c | 12 months
  This is a blood test of the patient.
Apoprotein B | 12 months
  This is a blood test of the patient.
Apoportein A1 | 12 months
  This is a blood test of the patient.
Lawton Index | 12 months
  This is to messure the activities of daily living of the patient.
SF-36 | 12 months
  This is to messure the quality of life of the patient.
SIS | 12 months
  This is to messure the quality of life of the patient.
Stroke Self Management Questionary | 12 months
  This is to messure the self management satisfaction of the patient.
Stroke Management Questionary | 12 months
  This is to messure the self management satisfaction of the patient.
Satisfaction Questionary | 12 months
  This is to messure the self management satisfaction of the patient.
Post Stroke Checklist | 12 months
  This is to messure the adherence to the treatment of the patient.
Pharmacological Accountability | 12 months
  This is to messure the adherence to the treatment of the patient.
Non Pharmacological Accountability | 12 months
  This is to messure the adherence to the treatment of the patient.
Stroke Recurrences | 12 months
  This is to messure the complications of the patient.
Number of Readmissions | 12 months
  This is to messure the complications of the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Cruces, Barakaldo, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: No